CLINICAL TRIAL: NCT02336789
Title: Proposal to Examine the Effect of Fecal Transplantation on Obesity.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Malnick, doctor, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0088-14-KMC
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Disorientation as to People, Time and Place
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): 250 ml of normal saline (sham transplantation).
  Interventions: Other: normal saline
- intervention (Active Comparator): 250 ml of diluted fecal material prepared from a screened donor
  Interventions: Other: fecal material

INTERVENTIONS:
Other: fecal material — . All patients will undergo a screening colonoscopy and will be allocated to receive either 250 ml of diluted fecal material prepared from a screened donor, or an equivalent volume of normal saline (sham transplantation).
  Arms: intervention
Other: normal saline — All patients will undergo a screening colonoscopy and will be allocated to receive either 250 ml of diluted fecal material prepared from a screened donor, or an equivalent volume of normal saline (sham transplantation).
  Arms: placebo

SUMMARY:
The investigators propose to transplant feces from thin, disease-free donors into obese patients undergoing colonoscopy for screening for colorectal carcinoma.

The investigators will obtain feces from healthy donors with a BMI of between 21-24. The investigators will perform colonoscopy on healthy patients with a BMI of 30-40 kg/m2 who have a clear indication for a screening examination.

All patients will undergo a screening colonoscopy and will be allocated to receive either 250 ml of diluted fecal material prepared from a screened donor, or an equivalent volume of normal saline (sham transplantation).

The patients will be reviewed at 1 3 6 and 12 months. At this time note will be made of their weight, BMI and waist circumference. In addition note will be made of their fasting glucose and lipid profile.

DETAILED DESCRIPTION:
We propose to transplant feces from thin, disease-free donors into obese patients undergoing colonoscopy for screening for colorectal carcinoma.

We will obtain feces from healthy donors with a BMI of between 21-24, in accordance with the Protocol that was approved by the Israel Ministry of Health. The stool sample will be prepared as detailed below :

We will perform colonoscopy on healthy patients with a BMI of 30-40 kg/m2 who have a clear indication for a screening examination. These will be people who are above the age of 50 who have not had a screening colonoscopy in the last 10 years, or those with a family history of carcinoma of the colon who are over the age of 40 years.

All patients will undergo a screening colonoscopy and will be allocated to receive either 250 ml of diluted fecal material prepared from a screened donor, or an equivalent volume of normal saline (sham transplantation). The material will be injected in the amount of 50 ml at five locations- the terminal ileum (or the cecum if the terminal ileum cannot be intubated), ascending colon, transverse colon, descending colon and sigmoid colon- during withdrawal of the colonoscope from the cecum. The stool will not be delivered to the endoscopy suite until the patient is sedated and only the endoscopist performing the procedure will know what treatment arm the patient is in.

In addition, all patients participating in the study will receive standard advice regarding weight loss and physical activity (at least 90 minutes of walking for week) from a staff dietitian.

Stool samples will be obtained from the donor( from the stool donated for transplantation) and the patients at baseline (prior to transplantation), 1 month and 12 months and frozen at -80 C for high throughput analysis by standard techniques.

The patients will be reviewed at 1 3 6 and 12 months. At this time note will be made of their weight, BMI and waist circumference. In addition note will be made of their fasting glucose and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients with a BMI of 30-40 kg/m2 who have a clear indication for a screening examination. These will be people who are above the age of 50 who have not had a screening colonoscopy in the last 10 years, or those with a family history of carcinoma of the colon who are over the age of 40 years.

Exclusion Criteria:

* Exclusion criteria include hepatitis B and C infection,
* consumption of more than 20 gram of alcohol per day,
* diabetes mellitus treated with insulin,
* previous unstable coronary artery disease in the last year,
* HIV infection,
* concomitant use of corticosteroids in the previous 3 months and severe diverticulosis.

If patients were to receive antibiotic therapy during the year of follow up of the study, data will only be included in the analysis prior to this time.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
weight loss | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen DH Malnick, MD, Principal Investigator — Kaplan Medical Center; Ehud Melzer, MD, Study Director — Kaplan Medical Center
Locations (1):
- Kaplan Medical Center, Rehovot, Israel